CLINICAL TRIAL: NCT02863952
Title: Quantitation of Left Ventricular Ejection Fraction Change From Early Exercise Gated Stress/Rest Tc-99m CZT-SPECT MPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IORG0001472
Record Dates: First submitted 2016-07-24; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EARLY POST-STRESS EF CHANGE (Other): There is only a single arm. All patients undergoing the routine myocardial perfusion SPECT study will also have additional (earlier) image acquisition in order to assess the relation of early wall motion abnormalities to the severity of myocardial ischemia.
  Interventions: Other: Single photon emission computed tomography myocardial perfusion imaging; Device: novel cadmium-zinc-telluride (CZT) SPECT cameras

INTERVENTIONS:
Other: Single photon emission computed tomography myocardial perfusion imaging
Device: novel cadmium-zinc-telluride (CZT) SPECT cameras

SUMMARY:
The aim of this study is to evaluate early post-stress EF change (∆EF) and its relation to the severity of myocardial ischemia and angiographic coronary disease using CZT-SPECT MPI.

DETAILED DESCRIPTION:
Single photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI) is a well-established noninvasive procedure for the evaluation and risk stratification of patients with coronary artery disease (CAD). However, it has been recognized that in certain patients SPECT MPI is unable to detect the presence of CAD or underestimates its extent. The fact that moderate to severe perfusion defects are noted in less than half of the patients with significant left main disease has stimulated studies to improve the diagnostic accuracy of SPECT MPI. These studies have analyzed post-stress parameters such as left ventricular (LV) ejection fraction (EF), wall motion abnormalities and transient LV dilation. However, these parameters were derived from data acquired using conventional Anger cameras as long as 60 minutes after stress tracer injection. Such delayed assessment may miss early ischemic stunning as a result of its rapid transient changes. However, with highly sensitive detectors and short lived tracers, the ability of PET MPI to measure EF during peak of stress has been reported. Similarly, the novel cadmium-zinc-telluride (CZT) SPECT cameras with solid state cardiac-focused detectors are significantly more sensitive than the conventional Anger scintillation cameras giving to SPECT the "PET-like" ability to image rapidly right after the stress test. The aim of this study is to evaluate early post-stress EF change (∆EF) and its relation to the severity of myocardial ischemia and angiographic coronary disease using CZT-SPECT MPI.

ELIGIBILITY:
Inclusion Criteria: the patients who will be able to complete exercise treadmill testing will be enrolled and analyzed.

-

Exclusion Criteria:

* severe aortic stenosis
* resting heart rate > 130 beats/min
* significant atrial or ventricular arrhythmia
* sepsis
* fever
* hemodialysis
* pregnancy

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
ischemia by SPECT | 15-30 minutes post stress
  severity of inducible / reversible perfusion abnormalities